CLINICAL TRIAL: NCT03952650
Title: Sanaria PfSPZ Challenge With Pyrimethamine or Chloroquine Chemoprophylaxis Vaccination (PfSPZ-CVac Approach): A Randomized Double Blind Placebo Controlled Phase I/II Trial to Determine Safety and Protective Efficacy Against Natural Plasmodium Falciparum Infection in Bancoumana and Surrounding Areas, Mali
Brief Title: Sanaria PfSPZ Challenge With Pyrimethamine or Chloroquine Chemoprophylaxis Vaccination (PfSPZ-CVac Approach): A Randomized Double Blind Placebo Controlled Phase I/II Trial to Determine Safety and Protective Efficacy Against Natural Plasmodium Falcipa...
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 999919099; 19-I-N099
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-07

CONDITIONS: Malaria
Keywords: Field; Immunity; Chemoprophylaxis with Sporozoites; Vaccine; Malaria-Experienced
MeSH Terms: conditions — Malaria | interventions — chloroquine diphosphate; Pyrimethamine; Artemether, Lumefantrine Drug Combination; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- 1a (Experimental): Receiving 400,000 PfSPZ with 75 mg pyrimethamine day 0 post PfSPZ
  Interventions: Biological: PfSPZ Challenge; Drug: Pyrimethamine; Drug: Coartem
- 1b (Experimental): Receiving 400,000 PfSPZ with 75 mg pyrimethamine day 0 post PfSPZ
  Interventions: Biological: PfSPZ Challenge; Drug: Pyrimethamine; Drug: Coartem
- 2a (Experimental): Receiving 400,000 PfSPZ with 75 mg pyrimethamine days 2&3 post PfSPZ
  Interventions: Biological: PfSPZ Challenge; Drug: Pyrimethamine; Drug: Coartem
- 2b (Experimental): Receiving 400,000 PfSPZ with 75 mg pyrimethamine days 2&3 post PfSPZ
  Interventions: Biological: PfSPZ Challenge; Drug: Pyrimethamine; Drug: Coartem
- 3a (Experimental): Receiving 400,000 PfSPZ with chloroquine 2 days prior + 5 days post PfSPZibuprofen (if necessary)
  Interventions: Drug: Chloroquine Phosphate; Biological: PfSPZ Challenge; Drug: Coartem; Drug: ibuprofen
- 3b (Experimental): Receiving 400,000 PfSPZ with weekly chloroquineibuprofen (if necessary)
  Interventions: Drug: Chloroquine Phosphate; Biological: PfSPZ Challenge; Drug: Coartem; Drug: ibuprofen
- 4a (Placebo Comparator): Receiving normal saline with 75 mg pyrimethamine day 0 post injection
  Interventions: Drug: Pyrimethamine; Drug: Coartem
- 4b (Placebo Comparator): Receiving normal saline with 75 mg pyrimethamine days 2&3 post injection
  Interventions: Drug: Pyrimethamine; Drug: Coartem
- 4c (Placebo Comparator): Receiving normal saline with weekly chloroquineibuprofen (if necessary)
  Interventions: Drug: Chloroquine Phosphate; Drug: Coartem; Drug: ibuprofen
- 5a (Experimental): Receiving 300,000 PfSPZ with 75 mg pyrimethamine day 0 post PfSPZ (if necessary)
  Interventions: Biological: PfSPZ Challenge; Drug: Pyrimethamine; Drug: Coartem
- 5b (Experimental): Receiving 300,000 PfSPZ with 75 mg pyrimethamine day 0 post PfSPZ
  Interventions: Biological: PfSPZ Challenge; Drug: Pyrimethamine; Drug: Coartem
- 6a (Experimental): Receiving 300,000 PfSPZ with 75 mg pyrimethamine days 2&3 post PfSPZ (if necessary)
  Interventions: Biological: PfSPZ Challenge; Drug: Pyrimethamine; Drug: Coartem
- 6b (Experimental): Receiving 300,000 PfSPZ with 75 mg pyrimethamine days 2&3 post PfSPZ (if necessary)
  Interventions: Biological: PfSPZ Challenge; Drug: Pyrimethamine; Drug: Coartem

INTERVENTIONS:
Drug: Chloroquine Phosphate — Chloroquine phosphate is approved for suppressive treatment (prophylaxis) and for acute attacks of malaria due to P. vivax, P. malariae, P. ovale, and susceptible strains of Pf. Chloroquine is a blood-stage schizonticide, highly active against replicating forms of blood-stage drug- sensitive parasites. As such, it is routinely employed as first-line prophylaxis against development of patent parasitemia and clinical malaria in non-immune travelers to areas with chloroquine sensitive Pf. In the pilot, chloroquine administration will begin with a loading dose 2 days prior to PfSPZ Challenge and finishing with a maintenance dose 5 days after PfSPZ Challenge. In the main phase, chloroquine will be first administered as a loading dose 2 days prior to PfSPZ Challenge and continuing weekly using a maintenance dose for a total of 10 doses, finishing with a last dose 5 days after the third injection with PfSPZ Challenge.
  Arms: 3a; 3b; 4c
Biological: PfSPZ Challenge — PfSPZ Challenge (NF54) acts as the immunogen in the PfSPZ-CVac approach to vaccinating against malaria. Participants will receive either one (in the pilot phase) or 3 (in the main phase) 400,000 or 300,000 aseptic, purified, cryopreserved, fully infectious PfSPZ injections by DVI (with concurrent administration of antimalarial drugs). Following immunization, participants in the main phase will be followed through the transmission season in order to assess vaccine efficacy.
  Arms: 1a; 1b; 2a; 2b; 3a; 3b; 5a; 5b; 6a; 6b
Drug: Pyrimethamine — Pyrimethamine has been FDA approved for acute treatment and chemoprophylaxis of malaria due to susceptible strains of plasmodia.
  Pyrimethamine has been shown to possess both liver and blood stage activity. In this study, we plan to use a higher dose of pyrimethamine, 75 mg orally for either one or two days each month. The pilot arms will receive either a total of 1 daily dose or 2 daily doses. The main arms will receive a total of 3 daily doses or a total of 6 doses.
  Arms: 1a; 1b; 2a; 2b; 4a; 4b; 5a; 5b; 6a; 6b
Drug: Coartem — Antimalarial (Coartem ) will be administered to all participants twice during the study, approximately 2 weeks prior to the first vaccination in order to clear pre-existing parasitemia that may interfere with immunity development. The second dose will be given approximately 2 weeks prior to the 3rd vaccination in order to clear any parasitemia infection that may have happened naturally during the vaccination period and prior to the follow up period.
Drug: ibuprofen — Ibuprofen likewise is not a part of the investigational product/regimen, but will be provided to participants in the chloroquine arm (Arm 4) if required to mitigate typical symptoms of malaria infection such as headache, myalgia, fever and chills.
  Arms: 3a; 3b; 4c

SUMMARY:
Background:

Malaria remains a major global health problem. Malaria is spread by the bite of mosquitos. Africa is the region of the world where most people get malaria. Sanaria PfSPZ Challenge is a malaria vaccine. Researchers want to see if the vaccine combined with partner drugs can help protect against malaria.

Objective:

To test if injections with 3 monthly doses of Sanaria PfSPZ Challenge, combined with either pyrimethamine (PYR) or chloroquine as a partner drug, is safe, tolerable, and effective.

Eligibility:

Healthy people ages 18-50 years who live in Bancoumana, Mali, or nearby

Design:

Participants will be screened with the Malaria Comprehension Exam to check their understanding of the study. They will have a medical history. They will have a physical exam. They will have blood tests, urine tests, and heart tests.

Participants will join either the pilot study or the main study.

Participants will be assigned to groups. Depending on their group, they will get at least one injection of either a placebo or the vaccine. They may have up to 3 vaccines, 4 weeks apart. The injection will be into a vein with a needle.

Participants will also take pyrimethamine or chloroquine by mouth. They will also take standard doses of antimalarial drugs by mouth.

Participants will have blood tests throughout the study.

Participants may develop a rash or injection site reaction. If this happens, photos of the site may be taken.

Participants will be observed for infection for many days after the injections.

DETAILED DESCRIPTION:
Human studies have shown that immunization by the bite of Plasmodium falciparum (Pf) sporozoite (SPZ)-infected mosquitoes (chemoprophylaxis with sporozoites [CPS]) or by injecting aseptic, purified, cryopreserved sporozoites (SPZ) with needle and syringe (PfSPZ chemoprophylaxis vaccination, Sanaria PfSPZ-CVac) under drug coverage with chloroquine can provide >80% protection against homologous controlled human malaria infection (CHMI) (Roestenberg, McCall et al. 2009, Roestenberg, Teirlinck et al. 2011, Mordmuller, Surat et al. 2017). The protective immunity induced by CPS/PfSPZ-CVac is thought to target sporozoite and liver stage antigens, but the transient parasitemia observed under chloroquine prophylaxis may additionally induce immune responses targeting blood stage parasites that contribute to protection. It is important to understand the contribution of each stage in this model as transient parasitemia in the immunization process adds a safety concern and may impair the development of immunity.

We have conducted two phase 1 studies to explore whether significant protective efficacy can be achieved with exclusively pre-erythrocytic (sporozoite/liver stage) exposure in this model using PYR chemoprophylaxis. This drug, unlike chloroquine, kills the parasites in the liver, so there is no period of transient parasitemia following immunization. These studies in malaria na(SqrRoot) ve adults demonstrated that PfSPZ-CVac (with PYR administered 2 & 3 days after injection) is safe, well-tolerated, and can prevent subpatent and patent parasitemia after PfSPZ injection. The NCT02511054 study used the same dose (5.12x104 PfSPZ) that has resulted in >80% protection in previous trials of PfSPZ-CVac (chloroquine), showed only 2/9 vaccinees were protected against a homologous (same strain of Pf as the vaccine) CHMI. In trials using irradiated SPZ, increasing the dose of PfSPZ used for immunization has resulted in higher protective efficacy. Therefore, in an ongoing trial, NCT03083847, we have increased the PfSPZ dose about 4-fold up to 2.0x105 PfSPZ, with preliminary results show markedly improved protection against both homologous and heterologous CHMI in healthy US adults (7/8 and 4/4 study subjects uninfected, respectively). This is the first demonstration that the PfSPZ-CVac approach can confer sterile protection without blood stage exposure.

Building on these promising results from PfSPZ-CVac (pyrimethamine) in the US, this proposed study in a malaria-endemic, adult population in Bancoumana, Mali will initially assess, in a pilot phase, the safety and tolerability of still higher doses of PfSPZ Challenge (4.0x105 PfSPZ) in combination with PYR (day 0;) or chloroquine (days -2, +5). The higher PfSPZ dose is hypothesized to be necessary to achieve significant efficacy against naturally transmitted malaria in malaria-experienced populations. Once this higher dose of PfSPZ is determined to be safe and tolerable and that earlier PYR dosing prevents patent parasitemia, the main phase will explore the effect of both earlier PYR dosing and a higher dosage of PfSPZ used for immunization in the development of protective immunity against natural malaria infection. The results of this study will contribute to understanding the targets and mechanisms of immunity against Pf malaria infection, and how the degree of prior exposure to the parasite (pre-erythrocytic and/or erythrocytic stages) impacts these responses and subsequent protective efficacy in field settings.

After completion of follow up in the main phase, all participants that are still enrolled in the study will be offered a booster dose of the vaccine (4th dose) with a single dose of 4x10^5 PfSPZ Challenge or normal saline (aligned with what they received in the main phase of the study) at approximately 11 months post 3rd vaccination. The booster dose is timed to allow administration well before the beginning of the ensuing malaria transmission season. Participants will then be followed for approximately 6 months to assess safety and vaccine efficacy through this second transmission season.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 and less than or equal to 50 years (for booster phase, age greater than or equal to 18 and less than or equal to 52 years)
* Resident of Bancoumana or nearby areas
* In good general health and without clinically significant medical history
* Malaria comprehension exam completed, passed (a score of greater than or equal to 80% or per investigator s discretion) and reviewed prior to enrollment
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
* Willing to have blood samples stored for future research
* Available for the duration of the study
* Females of childbearing potential must be willing to use reliable contraception (as defined below) from 21 days prior to first PfSPZ Challenge injection to 28 days following last PfSPZ Challenge exposure (or equivalent study day for Arm 5 controls). For the booster phase, this applies from 21 days prior to the booster vaccination to 28 days post booster vaccination.

  * Reliable methods of birth control include one of the following: confirmed pharmacologic contraceptives (parenteral) delivery; intrauterine or implantable device. OR
  * Reliable methods of birth control include concurrent use of a pharmacologic and a barrier method, i.e., two of the following: confirmed pharmacologic contraceptives (oral, transdermal) delivery or vaginal ring AND condoms with spermicide or diaphragm with spermicide. OR
  * Non-childbearing women will also be required to report date of last menstrual period, history of surgical sterility (i.e. tubal ligation, hysterectomy) or premature ovarian insufficiency (POI), and will have urine or serum pregnancy test performed per protocol.
* For booster phase only: previously or currently enrolled in protocol #19-I-N099 and completed all three primary vaccinations.

EXCLUSION CRITERIA:

* Pregnancy, as determined by a positive urine or serum human choriogonadotropin (beta-hCG) test (if female)

  --NOTE: Pregnancy is also a criterion for discontinuation of any further dosing or non-safety related interventions for that subject.
* Currently breast-feeding (if female)
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol
* Hemoglobin, WBC, absolute neutrophils, and platelets outside the local laboratorydefined limits of normal (subjects may be included at the investigator s discretion for 'not clinically significant' values)
* Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratoryMali PfSPZ-CVac (pyrimethamine) defined upper limit of normal (subjects may be included at the investigator s discretion for not clinically significant values)
* Infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B (HBV) (For the booster phase: re-testing NOT required for enrollment unless clinically indicated)
* Known or documented sickle cell disease by history (Note: known sickle cell trait is NOT exclusionary)
* Clinically significant abnormal electrocardiogram (ECG) (For the booster phase: re-testing NOT required for enrollment unless clinically indicated)
* Moderate or high risk for coronary heart disease (CHD) based on NHANES I cardiovascular risk assessment
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis
* History of receiving any other investigational product within the past 30 days
* Participation or planned participation in a clinical trial with an investigational product prior to completion of the last required protocol follow-up visit
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (defined as asthma that is unstable or required emergent care,urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years)
* Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sj(SqrRoot)(Delta)gren s syndrome, or autoimmune thrombocytopenia
* Known immunodeficiency syndrome
* Known asplenia or functional asplenia
* Use of:
* a. Chronic (greater than or equal to 14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of vaccination
* b. Antimalarials for example artemether, artemether-lumefantrine, artesunate, artesunate-amodiaquine, other than those prescribed by the investigator as part of the study procedures within 14 days prior to the first vaccine
* c. Systemic antibiotics with known antimalarial activity such as trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, ciprofloxacin or azithromycin within 5 half-lives of the drug prior to the first vaccine
* Receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks prior to Vaccination #1 and every subsequent vaccination day
* Receipt of immunoglobulins and/or blood products within the past 6 months
* Previous receipt of an investigational anti-infectivity malaria vaccine in the last 2 years (this requirement is waived for the booster phase)
* Known allergies or contraindication against: PYR, chloroquine, NSAIDs, artemether, lumefantrine
* Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Vaccine Center STTB/MRTC, Bamako, Mali

REFERENCES:
- [Background] Bijker EM, Borrmann S, Kappe SH, Mordmuller B, Sack BK, Khan SM. Novel approaches to whole sporozoite vaccination against malaria. Vaccine. 2015 Dec 22;33(52):7462-8. doi: 10.1016/j.vaccine.2015.09.095. Epub 2015 Oct 23. PMID 26469716
- [Background] Mordmuller B, Surat G, Lagler H, Chakravarty S, Ishizuka AS, Lalremruata A, Gmeiner M, Campo JJ, Esen M, Ruben AJ, Held J, Calle CL, Mengue JB, Gebru T, Ibanez J, Sulyok M, James ER, Billingsley PF, Natasha KC, Manoj A, Murshedkar T, Gunasekera A, Eappen AG, Li T, Stafford RE, Li M, Felgner PL, Seder RA, Richie TL, Sim BK, Hoffman SL, Kremsner PG. Sterile protection against human malaria by chemoattenuated PfSPZ vaccine. Nature. 2017 Feb 23;542(7642):445-449. doi: 10.1038/nature21060. Epub 2017 Feb 15. PMID 28199305
- [Background] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, enrollment occurs with receipt of the first dose of artemether/lumefantrine and collection of baseline study samples on study Day -17.
Groups:
- 1a - Pilot/Safety: Dosing Interval on Days: 1: Participants received 1 dose of 4x10^5 PfSPZ via direct venus inoculation (DVI) with 75 mg PYR day 0 post PfSPZ
- 1b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57: Participants received 4x10^5 PfSPZ via direct venus inoculation (DVI) with 75 mg PYR day 0 post PfSPZ on day 1, day 29 and day 57.
- 2a - Pilot/Safety: Dosing Interval on Days: 1: Participants received 1 dose of 4x10^5 PfSPZ via direct venus inoculation (DVI) with 75 mg PYR day 2 & 3 post PfSPZ
- 2b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57: Participants received 4x10^5 PfSPZ via direct venus inoculation (DVI) with 75 mg PYR day 2 & 3 post PfSPZ on day 1, day 29 and day 57.
- 3a - Pilot/Safety: Dosing Interval on Days: 1: Participants received 1 dose of 4x10^5 PfSPZ via direct venus inoculation (DVI) with chloroquine 2 days prior & 5 days post PfSPZ
- 4a - Safety Comparator: Dosing Interval on Days: 1, 29, 57: Participants received normal saline (NS) via direct venus inoculation (DVI) with 75 mg PYR day 0 post PfSPZ on day 1, day 29 and day 57.
- 4b - Safety Comparator: Dosing Interval on Days: 1, 29, 57: Participants received normal saline (NS) via direct venus inoculation (DVI) with 75 mg PYR day 2 & 3 post PfSPZ on day 1, day 29 and day 57.
Period: Overall Study
Arm/Group | 1a - Pilot/Safety: Dosing Interval on Days: 1 | 1b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 | 2a - Pilot/Safety: Dosing Interval on Days: 1 | 2b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 | 3a - Pilot/Safety: Dosing Interval on Days: 1 | 4a - Safety Comparator: Dosing Interval on Days: 1, 29, 57 | 4b - Safety Comparator: Dosing Interval on Days: 1, 29, 57
Started | 4 | 90 | 4 | 60 | 4 | 54 | 36
Completed | 4 | 83 | 4 | 53 | 4 | 47 | 32
Not Completed | 0 | 7 | 0 | 7 | 0 | 7 | 4
Not completed — TRAVEL | 0 | 4 | 0 | 4 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 3 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Received wrong vaccine and travelled | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Unable to make study visit | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1a - Pilot/Safety: Dosing Interval on Days: 1 | 1b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 | 2a - Pilot/Safety: Dosing Interval on Days: 1 | 2b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 | 3a - Pilot/Safety: Dosing Interval on Days: 1 | 4a - Safety Comparator: Dosing Interval on Days: 1, 29, 57 | 4b - Safety Comparator: Dosing Interval on Days: 1, 29, 57 | Total
Number analyzed (Participants) | 4 | 90 | 4 | 60 | 4 | 54 | 36 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 90 | 4 | 60 | 4 | 54 | 36 | 252
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (14.4) | 34.6 (10.0) | 23.8 (10.8) | 34.5 (10.0) | 31.8 (10.9) | 34.6 (10.0) | 34.9 (9.9) | 34.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 27 | 0 | 21 | 3 | 19 | 12 | 84
  Male | 2 | 63 | 4 | 39 | 1 | 35 | 24 | 168
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Malinke | 3 | 74 | 3 | 53 | 4 | 48 | 30 | 215
  Bozo | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Bambara | 0 | 3 | 0 | 3 | 0 | 3 | 2 | 11
  Bobo | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Minianka | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3
  Peulh | 0 | 8 | 0 | 3 | 0 | 2 | 4 | 17
  Sarakole | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Sonrhai | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Mali | 4 | 90 | 4 | 60 | 4 | 54 | 36 | 252

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Sensitive Blood Smear (sBS)
Description: Count of participants with positive sensitive blood smear (sBS) occurring after PfSPZ-CVac immunization starting on day 7 post DVI. Only pilot phase arms (Arms 1a, 2a) were analyzed for this outcome measure. Arms 5a and 6a were not performed, as no patent parasitemia was observed in either Arms 1a or 2a, per the protocol.
Time Frame: 7 -12 days post-inoculation
Measure: Count of Participants; unit: Participants
Arm/Group | 1a - Pilot/Safety: Dosing Interval on Days: 1 | 2a - Pilot/Safety: Dosing Interval on Days: 1
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Local and Systemic Grade 3 Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Count of participants with local and systemic grade 3 signs or symptoms lasting more than 48 hours despite adequate management and serious adverse events (SAEs) occurring after PfSPZ-CVac DVI. Only arm 3a was analyzed for this outcome measure, per the protocol objectives.
Time Frame: From day of inoculation to 14 days post-inoculation
Measure: Count of Participants; unit: Participants
Arm/Group | 3a - Pilot/Safety: Dosing Interval on Days: 1
Number analyzed (Participants) | 4
Participants | 0

3. Primary Outcome: Number of Participants With Local and Systemic Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Count of participants with local and systemic adverse events (AEs) and serious adverse events (SAEs) occurring after PfSPZ-CVac immunization. This outcome measure applies to main phase arms 1b, 2b, 4a, and 4b. Arms 5b and 6b were not performed as patent parasitemia with the higher dose of PfSPZ was not observed in the pilot phase (Arms 1a, 2a).
Time Frame: For the main phase: from the day of inoculation to approximately 6 months post-3rd inoculation. For the booster phase: from the time of inoculation to approximately 6 months post-booster inoculation
Measure: Count of Participants; unit: Participants
Arm/Group | 1b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 | 2b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 | 4a - Safety Comparator: Dosing Interval on Days: 1, 29, 57 | 4b - Safety Comparator: Dosing Interval on Days: 1, 29, 57
Number analyzed (Participants) | 90 | 60 | 54 | 36
Participants | 88 | 59 | 51 | 36

ADVERSE EVENTS:
Time Frame: One month for pilot phase; eight months for main phase; seven months for booster phase
Arm/Group | 1a - Pilot/Safety: Dosing Interval on Days: 1 | 1b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 | 2a - Pilot/Safety: Dosing Interval on Days: 1 | 2b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 | 3a - Pilot/Safety: Dosing Interval on Days: 1 | 4a - Safety Comparator: Dosing Interval on Days: 1, 29, 57 | 4b - Safety Comparator: Dosing Interval on Days: 1, 29, 57
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/90 | 0/4 | 0/60 | 0/4 | 0/54 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/90 | 0/4 | 0/60 | 0/4 | 1/54 | 0/36
Other Adverse Events (participants affected / at risk) | 1/4 | 88/90 | 1/4 | 59/60 | 2/4 | 51/54 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1a - Pilot/Safety: Dosing Interval on Days: 1 (N=4) | 1b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 (N=90) | 2a - Pilot/Safety: Dosing Interval on Days: 1 (N=4) | 2b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 (N=60) | 3a - Pilot/Safety: Dosing Interval on Days: 1 (N=4) | 4a - Safety Comparator: Dosing Interval on Days: 1, 29, 57 (N=54) | 4b - Safety Comparator: Dosing Interval on Days: 1, 29, 57 (N=36)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1a - Pilot/Safety: Dosing Interval on Days: 1 (N=4) | 1b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 (N=90) | 2a - Pilot/Safety: Dosing Interval on Days: 1 (N=4) | 2b - Safety/Efficacy: Dosing Interval on Days: 1, 29, 57 (N=60) | 3a - Pilot/Safety: Dosing Interval on Days: 1 (N=4) | 4a - Safety Comparator: Dosing Interval on Days: 1, 29, 57 (N=54) | 4b - Safety Comparator: Dosing Interval on Days: 1, 29, 57 (N=36)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 8 (8) | 0 (0) | 1 (1) | 4 (5)
Blood creatinine increased (Investigations) | 0 (0) | 38 (83) | 1 (1) | 27 (55) | 0 (0) | 17 (30) | 17 (27)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 7 (7) | 0 (0) | 2 (2) | 0 (0) | 7 (9) | 2 (2)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 9 (9) | 0 (0) | 7 (7) | 0 (0) | 14 (15) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 15 (18) | 0 (0) | 8 (11) | 1 (1) | 16 (17) | 3 (8)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye burns (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 10 (12) | 0 (0) | 7 (8) | 0 (0) | 9 (13) | 4 (7)
Gastroenteritis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 4 (5) | 6 (6)
Genital infection (Infections and infestations) | 0 (0) | 6 (6) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 27 (36) | 0 (0) | 24 (34) | 0 (0) | 24 (37) | 19 (30)
Hemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 7 (8) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 40 (85) | 0 (0) | 24 (50) | 0 (0) | 12 (23) | 13 (31)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 30 (40) | 0 (0) | 24 (31) | 0 (0) | 32 (42) | 19 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 36 (71) | 0 (0) | 14 (32) | 0 (0) | 11 (21) | 11 (26)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 3 (4) | 5 (7)
Otitis media (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 10 (12) | 0 (0) | 5 (8) | 0 (0) | 4 (5) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 48 (92) | 0 (0) | 38 (68) | 1 (1) | 27 (47) | 22 (42)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinobronchitis (Infections and infestations) | 0 (0) | 9 (9) | 0 (0) | 7 (7) | 0 (0) | 9 (12) | 4 (4)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 6 (6) | 0 (0) | 2 (2) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 11 (11) | 0 (0) | 9 (12) | 0 (0) | 9 (11) | 4 (6)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT03952650/Prot_SAP_000.pdf